CLINICAL TRIAL: NCT05137613
Title: One and Two-visit Root Canal Retreatment in Teeth With Periapical Lesion
Brief Title: One and Two-visit Root Canal Retreatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Seniha Miçooğulları Kurt, Asst. Assoc. Dr, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Root canal retreatment
Record Dates: First submitted 2021-11-17; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Root Canal Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One visit root canal retreatment (Active Comparator): The teeth were treated in one-visit (OV) root canal retreatment. Final root canal irrigation was performed with 5% EDTA, followed by 2.5% NaOCl and received an additional final rinse with 2% CHX before obturation.
  Interventions: Other: One visit root canal retreatment
- Two visit root canal retreatment (Active Comparator): The teeth were treated in two visit (TV) root canal retreatment. After completion of root canal instrumentation, calcium hydroxide (CH) paste was placed into the root canal. In second visit, all root canals were irrigated with 5% EDTA followed by 2.5% NaOCl before obturation.
  Interventions: Other: Two visit root canal retreatment

INTERVENTIONS:
Other: One visit root canal retreatment — The teeth were treated in one-visit (OV) root canal retreatment. Final root canal irrigation was performed with 5% EDTA, followed by 2.5% NaOCl and received an additional final rinse with 2% CHX before obturation
  Arms: One visit root canal retreatment
Other: Two visit root canal retreatment — The teeth were treated in two visit (TV) root canal retreatment. After completion of root canal instrumentation, calcium hydroxide (CH) paste was placed into the root canal. In second visit, all root canals were irrigated with 5% EDTA followed by 2.5% NaOCl before obturation.
  Arms: Two visit root canal retreatment

SUMMARY:
A hundred previously root canal treated asymptomatic single-rooted teeth with periapical lesions were treated in single versus multiple visit root canal retreatment. Half of the teeth were randomly assigned to the one-visit (OV) group. The other teeth were treated in two visits (TV). All patients were recalled and investigated clinically and radiographically for 24 months.

DETAILED DESCRIPTION:
The aim of the study was to evaluate the radiographic evidence of periapical healing in previously root canal treated teeth with apical periodontitis treated in a single visit and to compare the results with conventional two-visit root canal treatment .100 asymptomatic single rooted teeth with periapical lesions were included. The root canal filling material was removed and reinstrumentation was performed using hand files with 2.5% sodium hypochlorite (NaOCl) and 5% ethylenediaminetetraacetic acid (EDTA) as irrigants. Half of the teeth were randomly assigned to the one-visit (OV) group. The other teeth were treated in two visits (TV), after completion of root canal instrumentation calcium hydroxide paste was placed into the root canal and root canal obturation was performed in second visit. All patients were recalled and investigated clinically and radiographically for 24 months. Changes in apical bone density indicating radiographic healing were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* with a non-contributory medical history,
* single-rooted teeth with periapical lesions,
* previously root canal treated but no reduction in the lesion after the treatment
* diagnosed as asymptomatic apical periodontitis

Exclusion Criteria:

* clinical symptoms, drainage,
* more than 5 mm loss of periodontal attachment,
* non-restorable tooth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
The presence or absence of clinical symptoms in clinical examination | 24 months
  All patients were called for follow up visits. The evaluation was performed by clinical examination. Clinical symptoms including presence of pain, tenderness to percussion and palpation, presence of sinus tract or swelling was detected and recorded as present or absent. If one of these symptoms recorded as present, it is considered as failure. If there is no symptom, it is considered as success.
The rate of radiographic healing of the periapical lesion. | 24 months
  Follow-up visits were performed for all patients in order to evaluate radiographic status. Changes in apical bone density indicating radiographic healing was assessed using Periapical Index (PAI) (Orstavik 1986) as the scoring system. PAI 1 and 2 considered as healed, reduction in the PAI score was considered as healing and persistence or increased in the PAI score (PAI 4 or 5) was considered as failure.

SECONDARY OUTCOMES:
The level of postoperative pain | 12hours-24hours and 48 hours
  Postoperative pain after 12, 24 and 48 hours, was measured using a modified 4-grade visual analogue scale (VAS) ranging from 1 (no pain), 2 (mild pain), 3 (moderate pain/pain relieved by analgesics), to 4 (severe pain).

CONTACTS AND LOCATIONS:
Overall Officials: Fulya Karaoglan, Principal Investigator — Ege University Faculty of Dentistry
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eyuboglu TF, Olcay K, Ozcan M. A clinical study on single-visit root canal retreatments on consecutive 173 patients: frequency of periapical complications and clinical success rate. Clin Oral Investig. 2017 Jun;21(5):1761-1768. doi: 10.1007/s00784-016-1957-2. Epub 2016 Sep 22. PMID 27660159
- [Background] He J, White RK, White CA, Schweitzer JL, Woodmansey KF. Clinical and Patient-centered Outcomes of Nonsurgical Root Canal Retreatment in First Molars Using Contemporary Techniques. J Endod. 2017 Feb;43(2):231-237. doi: 10.1016/j.joen.2016.10.029. PMID 28132709
- [Background] Zhang MM, Fang GF, Chen XT, Liang YH. Four-year Outcome of Nonsurgical Root Canal Retreatment Using Cone-beam Computed Tomography: A Prospective Cohort Study. J Endod. 2021 Mar;47(3):382-390. doi: 10.1016/j.joen.2020.10.020. Epub 2020 Oct 29. PMID 33130061